CLINICAL TRIAL: NCT02736487
Title: Effect of Short-term Portable Air Purifier Use on Occupant Health Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Duke University (Other); Tsinghua University (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, Feng Li, MD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2015[38]
Record Dates: First submitted 2015-12-10; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Non-smoking, Healthy Adults
Keywords: Air Pollution; Exposure Assessment; Filtration; Cardiovascular Outcomes; Respiratory Outcomes; Short-term Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: True-Washout-Sham (Active Comparator): Subjects in group A receives true air filtration intervention, then at least two weeks of washout period, followed by sham air filtration intervention.
  Interventions: Device: True-Washout-Sham Air Filtration Intervention
- Group B: Sham-Washout-True (Active Comparator): Subjects in group B receives sham air filtration intervention, then at least two weeks of washout period, followed by true air filtration intervention.
  Interventions: Device: Sham-Washout-True Air Filtration Intervention

INTERVENTIONS:
Device: True-Washout-Sham Air Filtration Intervention — This intervention involved three sequential steps: (1) 12 to 20 hours of true air filtration intervention; (2) at least two weeks of washout period; (3) 12 to 20 hours of sham air filtration intervention. In the indoor environment, the portable filtration device drew room air, sent it through filter and active carbon (for true filtration) or active carbon alone (sham filtration) and then delivered processed air back to room air. In the study the portable filtration device processes 2.8 cubic meter of room air per minute. The washout period lasted for at least two weeks where no filtration intervention was implemented.
  Arms: Group A: True-Washout-Sham
Device: Sham-Washout-True Air Filtration Intervention — This intervention involved three sequential steps: (1) 12 to 20 hours of sham air filtration intervention; (2) at least two weeks of washout period; (3) 12 to 20 hours of true air filtration intervention. In the indoor environment, the portable filtration device drew room air, sent it through filter and active carbon (for true filtration) or active carbon alone (sham filtration) and then delivered processed air back to room air. In the study the portable filtration device processes 2.8 cubic meter of room air per minute. The washout period lasted for at least two weeks where no filtration intervention was implemented.
  Arms: Group B: Sham-Washout-True

SUMMARY:
The purpose of this research project is to examine whether short-term use of portable air pollution filtration can result in changes in indoor airborne pollutants and impact on cardiovascular and respiratory health outcomes of the inhabitants.

DETAILED DESCRIPTION:
This study will focus on evaluating the short-term benefits of a common portable air purifier technology in reducing air pollutant exposure and the anticipated concomitant health impacts. High ambient levels of various air pollutants in the Shanghai area serve as a useful model to test the portable air purifier intervention in a realistic setting. As most people using a portable air purifier would only be able to do so in their residences, the investigators have designed our study only to test residential air purifier use. Our hypothesis is that the reduction in pollutant concentrations in indoor air caused by the air purifier will result in measurable reductions in risk factors for cardiovascular and respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking adults
* Live in the dormitory building at Shanghai First People's Hospital (South Section).

Exclusion Criteria:

* Current smokers
* Has any of the following diseases: chronic respiratory, cardiovascular, liver, renal, hematological disease; diabetes mellitus;
* Has any other diseases that may confound or complicate the effects of the intervention
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline FEV1 (forced expiratory volume in the first second of exhalation) within 2h after the filtration intervention | Within 2h after the filtration intervention
  FEV1 (forced expiratory volume in the first second of exhalation, unit: liter) was measured by spirometry in all subjects within 2h after the filtration intervention to compare to FEV1 value of study subjects at baseline (i.e. at start of the study).
Change from baseline R5 (airway resistance measured at 5Hz) within 2h after the filtration intervention | Within 2h after the filtration intervention
  R5 (airway resistance measured at 5Hz) was accessed by impulse oscillometry in all subjects within 2h after the filtration intervention to compare to the R5 value of study subjects at baseline (i.e. before the start of intervention).
Change in baseline exhaled nitric oxide (eNO) within 2h after the filtration intervention | Within 2h after the filtration intervention
  Exhaled nitric oxide (eNO) was measured in all subjects within 2h after the filtration intervention to compare to the exhaled nitric oxide measurement of study subjects at baseline (i.e. before the start of intervention). Exhaled breath is collected in air sampling bags, and the concentration of NO was quantified by Thermo Scientific model 42i (NO-NO2-NOx) analyzer.
Change in exhaled nitric oxide (eNO) at 6h after filtration intervention compared to baseline | 6h after filtration intervention
  Exhaled nitric oxide (eNO) was measured in all subjects 6h after filtration intervention to compare to the exhaled nitric oxide measurement of study subjects at baseline (i.e. before the start of intervention). Exhaled breath is collected in air sampling bags, and the concentration of NO was quantified by Thermo Scientific model 42i (NO-NO2-NOx) analyzer.
Change from baseline PWV (pulse wave velocity) within 2h after the filtration intervention | Within 2h after the filtration intervention
  PWV (pulse wave velocity) was measured by the VICORDER instrument in all subjects right after filtration intervention to compare to the PWV value measured at baseline (i.e. before the start of intervention).

SECONDARY OUTCOMES:
Change from baseline urinary biomarkers of inflammation and oxidative stress at 0h after the filtration intervention | At 0h after the filtration intervention
  Urine samples were collected from each subject at 0h after the filtration intervention to quantify changes in urinary oxidative stress and inflammation biomarkers compared to baseline (i.e. before intervention). The urinary biomarkers to be analyzed include: malondialdehyde (MDA), 8-hydroxy-2' -deoxyguanosine (8-OHdG) and creatinine. The unit of the urinary biomarkers will be reported as micro molar/ milliliter.
Change in baseline urinary biomarkers of inflammation and oxidative stress at 6h after filtration intervention | 6h after filtration intervention
  Urine samples were collected from each subject at 6h after filtration intervention to quantify changes in urinary oxidative stress and inflammation biomarkers compared to baseline (i.e. before intervention). The urinary biomarkers to be analyzed include: malondialdehyde (MDA), 8-hydroxy-2' -deoxyguanosine (8-OHdG) and creatinine. The unit of the urinary biomarkers will be reported as micro molar/ milliliter.
Change in baseline urinary biomarkers of inflammation and oxidative stress at 24h after filtration intervention | 24h after filtration intervention
  Urine samples were collected from each subject at 24h after filtration intervention to quantify changes in urinary oxidative stress and inflammation biomarkers compared to baseline (i.e. before intervention). The urinary biomarkers to be analyzed include: malondialdehyde (MDA), 8-hydroxy-2' -deoxyguanosine (8-OHdG) and creatinine. The unit of the urinary biomarkers will be reported as micro molar/ milliliter.
Changes in baseline blood biomarkers of inflammation, oxidative stress and coagulation within 1h after filtration intervention | Within 1h after filtration intervention
  Blood samples were collected within 1h after filtration intervention for comparison of inflammatory and oxidative stress biomarkers to their baseline level (i.e. before the start of filtration intervention). Blood biomarkers that will be analyzed include: P-selectin, c-reactive protein, Von Willebrand factor and fibrinogen. The unit of the blood biomarkers will be reported as micro molar/ milliliter.
Changes in baseline blood biomarkers of inflammation, oxidative stress and coagulation right after filtration intervention | 24h after filtration intervention
  Blood samples were collected 24h after filtration intervention for comparison of inflammatory and oxidative stress biomarkers to their baseline level (i.e. before the start of filtration intervention). Blood biomarkers that will be analyzed include: P-selectin, c-reactive protein, Von Willebrand factor and fibrinogen. The unit of the blood biomarkers will be reported as micro molar/ milliliter.
Change in the duration of deep sleep on the first night and the second night of study participation | On the first night and the second night of study participation
  Duration of deep sleep was monitored by a sensor in a wristband on the first night and the second night of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Zhang, PhD, Principal Investigator — Duke University; Yinping Zhang, PhD, Principal Investigator — Tsinghua University
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided